CLINICAL TRIAL: NCT01476813
Title: A Randomized, Double-blind, Active-controlled, Cross-over Study to Assess Efficacy and Safety of 3 Free Doses of Glycopyrrolate With Beclomethasone/Formoterol pMDI for the Treatment of COPD Patients
Brief Title: Randomized Cross Over Study to Assess Efficacy and Safety of BDP/FF and Glycopyrrolate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1106-PR-0066
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glyco 25 (Experimental): BDP/FF (400/24 daily)+ Glyco 25µg daily
  Interventions: Drug: Glycopyrrolate
- Glyco 50 (Experimental): BDP/FF (400/24 daily)+ Glyco 50 µg daily
  Interventions: Drug: Glycopyrrolate
- Glyco 100 (Experimental): BDP/FF (400/24 daily)+ Glyco 100µg daily
  Interventions: Drug: Glycopyrrolate
- BDP/FF 400/24 (Active Comparator): BDP/FF 400/24
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: Glycopyrrolate — comparison of different dosages of drug
  Other Names: Foster+GLyco 25
  Arms: Glyco 25
Drug: Glycopyrrolate — comparison of different dosages of drug
  Other Names: Foster+GLyco 50
  Arms: Glyco 50
Drug: Glycopyrrolate — comparison of different dosages of drug
  Other Names: Foster+GLyco 100
  Arms: Glyco 100
Drug: Comparator — comparison of different dosages of drug versus comparator
  Other Names: Foster
  Arms: BDP/FF 400/24

SUMMARY:
dose-finding study to assess the optimal dose of glycopyrrolate daily dose on top of BDP/FF in COPD patients.

DETAILED DESCRIPTION:
A MULTICENTRE, RANDOMISED, DOUBLE-BLIND, ACTIVE-CONTROLLED, 4-WAY CROSS-OVER STUDY TO EVALUATE THE EFFICACY AND SAFETY OF A FREE COMBINATION OF 3 DOSES OF GLYCOPYRROLATE WITH FIXED COMBINATION BECLOMETHASONE DIPROPIONATE PLUS FORMOTEROL (FOSTER®) IN A METERED DOSE INHALER FOR THE TREATMENT OF PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE (COPD)

ELIGIBILITY:
Inclusion Criteria:

* COPD over 40 years of age (30 to 60% post-bronchodilator FEV1 predictive value)
* Patients under Double
* Patients under triple therapy (for 1 Mo prior Screening)

Exclusion Criteria:

* Pregnant or lactating women
* Patients experiencing a COPD exacerbation requiring use of systemic steroids and/or antibiotics, hospitalization
* concommitant diseases impacting feasibility or safety

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Aera under curve FEV1 AUC 0-12h | day 1 and 7 of treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Clinical Pharmacology and Respiratory Medicine, Medicines Evaluation Unit Ltd, Manchester University
Locations (1):
- Medicines Evaluation Unit Ltd., Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Result] Singh D, Schroder-Babo W, Cohuet G, Muraro A, Bonnet-Gonod F, Petruzzelli S, Hoffmann M, Siergiejko Z; TRIDENT study investigators. The bronchodilator effects of extrafine glycopyrronium added to combination treatment with beclometasone dipropionate plus formoterol in COPD: A randomised crossover study (the TRIDENT study). Respir Med. 2016 May;114:84-90. doi: 10.1016/j.rmed.2016.03.018. Epub 2016 Mar 26. PMID 27109816
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-003588-31
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-1106-PR-0066.pdf